CLINICAL TRIAL: NCT03843866
Title: The Use of Absorbable Suture Versus Tissue Glue in Laparoscopic Port Skin Closure. A Prospective, Randomised Control Trial. The STILS Trial.
Brief Title: Sutures Versus Glue in Laparoscopic Port Site Closure.
Acronym: STILS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Noel Edward Donlon, General Surgery Specialist Registrar, St. James's Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SJH 2019-1.0
Record Dates: First submitted 2019-02-12; First posted 2019-02-18 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Cosmetic Outcome; Infection; Cost
MeSH Terms: conditions — Infections | interventions — Sutures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suture & steri-strips (Active Comparator)
  Interventions: Other: 4-0 Monocryl
- Adhesive Glue (Active Comparator)
  Interventions: Other: Adhesive Glue

INTERVENTIONS:
Other: 4-0 Monocryl — sutures and steri-strips
  Other Names: sutures and steri strips
  Arms: Suture & steri-strips
Other: Adhesive Glue — Adhesive Glue
  Arms: Adhesive Glue

SUMMARY:
Cosmesis postoperatively is an important consideration for both patients and surgeons and consequently surgeons have become increasingly interested in replacing conventional sutures by means of adhesive bonds for the closure of skin wounds.

Therefore the investigators are using two different close techniques for laparoscopic wounds. These are; 1. sutures with steri-strips and 2. adhesive bond.

ELIGIBILITY:
Inclusion Criteria:

* Elective Laparoscopic surgeries. Emergency Laparoscopic surgeries.

Exclusion Criteria:

* Contaminated wounds. immunocompromised patients. diabetic patients. history of Keloid scarring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-09-02 (Estimated)

PRIMARY OUTCOMES:
Cosmesis | 6 months
  Cosmetic outcome being graded by patient and clinician via questionnaire. Observer scar assessment form (1-10) 1 = worst result possible, 10 being the best result possible.

SECONDARY OUTCOMES:
Surgical site infection (SSI). | 6 months
  Any superficial site infection which requires antibiotic use or wound complication such as dehisence. This information will be obtained from clinic.

CONTACTS AND LOCATIONS:
Locations (1):
- St. James Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramjit SE, Davey MG, Keelan S, Herlihy E, Dromey M, Garvey C, Nugent TS, Fawaz A, O'Connell L, Cunningham M, Fahy M, Ryan EJ, Moran B, Aljohmani L, Narayanasamy J, Kelly ME, Healy C, Donohoe C, Ravi N, Neary P, Reynolds JV, Donlon NE. Evaluating the use of absorbable sutures versus sTaples versus tIssue glue in laparoscopic port skin closure (STILS) trial: A prospective, multi-centre randomised clinical trial (RCT). Surgeon. 2025 Oct;23(5):306-312. doi: 10.1016/j.surge.2025.02.015. Epub 2025 Mar 17. PMID 40102141